CLINICAL TRIAL: NCT01221168
Title: ProGene: Etude Genetique et Epidemiologique du Cancer de la Prostate Familial
Brief Title: Epidemiologic and Genetic Study on Familial Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Centre de Recherche sur les Pathologies Prostatiques (Other)
Responsible Party: Sponsor
Other Study IDs: ProGene
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; genetic; epidemiology; susceptibility
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Disease Susceptibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from blood/saliva or urine Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Men with or without Prostate Cancer: Men with a histological confirmed prostate cancer, and their family members in case of hereditary prostate cancer.
  Men with no prostate cancer after a screening procedure for this disease, so that their biological samples can be compared to those of men with prostate cancer.

SUMMARY:
The aims of the study are:

* to identify genetic and molecular factors (rare mutations, polymorphisms) involved in the natural history of prostate cancers and their response to treatment,
* to evaluate and deduce their medical applications for screening and therapeutic management of these tumors.

DETAILED DESCRIPTION:
The impact of genetic factors on the natural history of prostate cancer (PC) is shown schematically at two levels:

1. first, at the constitutional level with germline alterations. Family history is found in 20% of PC patients. Different clinical entities associated with different modes of inheritance, susceptibility mutations or polymorphisms, define different evolutionary patterns. Also, studies suggested that some genetic polymorphisms alter the response to some treatments (such as recurrence after prostatectomy or radiotherapy) or adverse effects of those above (such as toxicity of radiation therapy).
2. secondly, PC is characterized by the accumulation of genetic alterations (somatic alterations or acquired mutations). These changes contribute in varying degrees to the aggressiveness of the disease (such as early metastatic potential) and treatment failure (such as resistance to radiation or hormone resistance).

The purpose of this study is to establish a register, with a follow up of cohort type and a collection of biological samples:

* For men with known prostate cancer.
* For men with no prostate cancer after a screening procedure for this disease, so that their biological samples can be compared to those of men with prostate cancer.

The registry data and collected biological samples are used to identify genetic and molecular factors involved in susceptibility, genesis and evolution of prostate cancers.

ELIGIBILITY:
Inclusion Criteria:

* patient with a histological confirmed prostate cancer
* member of a hereditary prostate cancer family
* healthy control men without prostate cancer

Exclusion Criteria:

* Absence of signed informed consent
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with or without prostate cancer are recruited in different departments of urology or care centers in France.
  For hereditary prostate cancer, patients and their family members are referred by all urologists from France.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 1996-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Performance of genetic and molecular factors in predicting the risk of prostate cancer | 20 years
  Logistic regression and artificial neural networks will be used

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Cussenot, MD, Ph.D., Principal Investigator — Centre de Recherche sur les Pathologies Prostatiques
Locations (5):
- France (5):
  - Department of Urology, CHU Angers, Angers
  - Department of Urology, Hopital de la Cavale Blanche, Brest
  - Department of Urology, CHU Dijon, Dijon
  - Department of Urology, Hopital Pitié-Salpetriere, Paris
  - Department of Urology, Hopital Tenon, Paris

REFERENCES:
- [Background] Cussenot O, Timms KM, Perrot E, Blanchet P, Brureau L, Solimeno C, Fromont G, Comperat E, Cancel-Tassin G. Tumour-based Mutational Profiles Predict Visceral Metastasis Outcome and Early Death in Prostate Cancer Patients. Eur Urol Oncol. 2024 Jun;7(3):597-604. doi: 10.1016/j.euo.2023.12.003. Epub 2024 Jan 5. PMID 38182487
- [Background] Wang A, Shen J, Rodriguez AA, Saunders EJ, Chen F, Janivara R, Darst BF, Sheng X, Xu Y, Chou AJ, Benlloch S, Dadaev T, Brook MN, Plym A, Sahimi A, Hoffman TJ, Takahashi A, Matsuda K, Momozawa Y, Fujita M, Laisk T, Figueredo J, Muir K, Ito S, Liu X; Biobank Japan Project; Uchio Y, Kubo M, Kamatani Y, Lophatananon A, Wan P, Andrews C, Lori A, Choudhury PP, Schleutker J, Tammela TLJ, Sipeky C, Auvinen A, Giles GG, Southey MC, MacInnis RJ, Cybulski C, Wokolorczyk D, Lubinski J, Rentsch CT, Cho K, Mcmahon BH, Neal DE, Donovan JL, Hamdy FC, Martin RM, Nordestgaard BG, Nielsen SF, Weischer M, Bojesen SE, Roder A, Stroomberg HV, Batra J, Chambers S, Horvath L, Clements JA, Tilly W, Risbridger GP, Gronberg H, Aly M, Szulkin R, Eklund M, Nordstrom T, Pashayan N, Dunning AM, Ghoussaini M, Travis RC, Key TJ, Riboli E, Park JY, Sellers TA, Lin HY, Albanes D, Weinstein S, Cook MB, Mucci LA, Giovannucci E, Lindstrom S, Kraft P, Hunter DJ, Penney KL, Turman C, Tangen CM, Goodman PJ, Thompson IM Jr, Hamilton RJ, Fleshner NE, Finelli A, Parent ME, Stanford JL, Ostrander EA, Koutros S, Beane Freeman LE, Stampfer M, Wolk A, Hakansson N, Andriole GL, Hoover RN, Machiela MJ, Sorensen KD, Borre M, Blot WJ, Zheng W, Yeboah ED, Mensah JE, Lu YJ, Zhang HW, Feng N, Mao X, Wu Y, Zhao SC, Sun Z, Thibodeau SN, McDonnell SK, Schaid DJ, West CML, Barnett G, Maier C, Schnoeller T, Luedeke M, Kibel AS, Drake BF, Cussenot O, Cancel-Tassin G, Menegaux F, Truong T, Koudou YA, John EM, Grindedal EM, Maehle L, Khaw KT, Ingles SA, Stern MC, Vega A, Gomez-Caamano A, Fachal L, Rosenstein BS, Kerns SL, Ostrer H, Teixeira MR, Paulo P, Brandao A, Watya S, Lubwama A, Bensen JT, Butler EN, Mohler JL, Taylor JA, Kogevinas M, Dierssen-Sotos T, Castano-Vinyals G, Cannon-Albright L, Teerlink CC, Huff CD, Pilie P, Yu Y, Bohlender RJ, Gu J, Strom SS, Multigner L, Blanchet P, Brureau L, Kaneva R, Slavov C, Mitev V, Leach RJ, Brenner H, Chen X, Holleczek B, Schottker B, Klein EA, Hsing AW, Kittles RA, Murphy AB, Logothetis CJ, Kim J, Neuhausen SL, Steele L, Ding YC, Isaacs WB, Nemesure B, Hennis AJM, Carpten J, Pandha H, Michael A, De Ruyck K, De Meerleer G, Ost P, Xu J, Razack A, Lim J, Teo SH, Newcomb LF, Lin DW, Fowke JH, Neslund-Dudas CM, Rybicki BA, Gamulin M, Lessel D, Kulis T, Usmani N, Abraham A, Singhal S, Parliament M, Claessens F, Joniau S, Van den Broeck T, Gago-Dominguez M, Castelao JE, Martinez ME, Larkin S, Townsend PA, Aukim-Hastie C, Bush WS, Aldrich MC, Crawford DC, Srivastava S, Cullen J, Petrovics G, Casey G, Wang Y, Tettey Y, Lachance J, Tang W, Biritwum RB, Adjei AA, Tay E, Truelove A, Niwa S, Yamoah K, Govindasami K, Chokkalingam AP, Keaton JM, Hellwege JN, Clark PE, Jalloh M, Gueye SM, Niang L, Ogunbiyi O, Shittu O, Amodu O, Adebiyi AO, Aisuodionoe-Shadrach OI, Ajibola HO, Jamda MA, Oluwole OP, Nwegbu M, Adusei B, Mante S, Darkwa-Abrahams A, Diop H, Gundell SM, Roobol MJ, Jenster G, van Schaik RHN, Hu JJ, Sanderson M, Kachuri L, Varma R, McKean-Cowdin R, Torres M, Preuss MH, Loos RJF, Zawistowski M, Zollner S, Lu Z, Van Den Eeden SK, Easton DF, Ambs S, Edwards TL, Magi R, Rebbeck TR, Fritsche L, Chanock SJ, Berndt SI, Wiklund F, Nakagawa H, Witte JS, Gaziano JM, Justice AC, Mancuso N, Terao C, Eeles RA, Kote-Jarai Z, Madduri RK, Conti DV, Haiman CA. Characterizing prostate cancer risk through multi-ancestry genome-wide discovery of 187 novel risk variants. Nat Genet. 2023 Dec;55(12):2065-2074. doi: 10.1038/s41588-023-01534-4. Epub 2023 Nov 9. PMID 37945903
- [Background] Cussenot O, Cancel-Tassin G, Rao SR, Woodcock DJ, Lamb AD, Mills IG, Hamdy FC. Aligning germline and somatic mutations in prostate cancer. Are genetics changing practice? BJU Int. 2023 Nov;132(5):472-484. doi: 10.1111/bju.16120. Epub 2023 Jul 27. PMID 37410655
- [Background] Darst BF, Shen J, Madduri RK, Rodriguez AA, Xiao Y, Sheng X, Saunders EJ, Dadaev T, Brook MN, Hoffmann TJ, Muir K, Wan P, Le Marchand L, Wilkens L, Wang Y, Schleutker J, MacInnis RJ, Cybulski C, Neal DE, Nordestgaard BG, Nielsen SF, Batra J, Clements JA, Cancer BioResource AP, Gronberg H, Pashayan N, Travis RC, Park JY, Albanes D, Weinstein S, Mucci LA, Hunter DJ, Penney KL, Tangen CM, Hamilton RJ, Parent ME, Stanford JL, Koutros S, Wolk A, Sorensen KD, Blot WJ, Yeboah ED, Mensah JE, Lu YJ, Schaid DJ, Thibodeau SN, West CM, Maier C, Kibel AS, Cancel-Tassin G, Menegaux F, John EM, Grindedal EM, Khaw KT, Ingles SA, Vega A, Rosenstein BS, Teixeira MR; NC-LA PCaP Investigators; Kogevinas M, Cannon-Albright L, Huff C, Multigner L, Kaneva R, Leach RJ, Brenner H, Hsing AW, Kittles RA, Murphy AB, Logothetis CJ, Neuhausen SL, Isaacs WB, Nemesure B, Hennis AJ, Carpten J, Pandha H, De Ruyck K, Xu J, Razack A, Teo SH; Canary PASS Investigators; Newcomb LF, Fowke JH, Neslund-Dudas C, Rybicki BA, Gamulin M, Usmani N, Claessens F, Gago-Dominguez M, Castelao JE, Townsend PA, Crawford DC, Petrovics G, Casey G, Roobol MJ, Hu JF, Berndt SI, Van Den Eeden SK, Easton DF, Chanock SJ, Cook MB, Wiklund F, Witte JS, Eeles RA, Kote-Jarai Z, Watya S, Gaziano JM, Justice AC, Conti DV, Haiman CA. Evaluating approaches for constructing polygenic risk scores for prostate cancer in men of African and European ancestry. Am J Hum Genet. 2023 Jul 6;110(7):1200-1206. doi: 10.1016/j.ajhg.2023.05.010. Epub 2023 Jun 12. PMID 37311464
- [Background] Cussenot O, Renard-Penna R, Montagne S, Ondet V, Pilon A, Guechot J, Comperat E, Hamdy F, Lamb A, Cancel-Tassin G. Clinical performance of magnetic resonance imaging and biomarkers for prostate cancer diagnosis in men at high genetic risk. BJU Int. 2023 Jun;131(6):745-754. doi: 10.1111/bju.15968. Epub 2023 Feb 6. PMID 36648168
- [Background] Chen F, Madduri RK, Rodriguez AA, Darst BF, Chou A, Sheng X, Wang A, Shen J, Saunders EJ, Rhie SK, Bensen JT, Ingles SA, Kittles RA, Strom SS, Rybicki BA, Nemesure B, Isaacs WB, Stanford JL, Zheng W, Sanderson M, John EM, Park JY, Xu J, Wang Y, Berndt SI, Huff CD, Yeboah ED, Tettey Y, Lachance J, Tang W, Rentsch CT, Cho K, Mcmahon BH, Biritwum RB, Adjei AA, Tay E, Truelove A, Niwa S, Sellers TA, Yamoah K, Murphy AB, Crawford DC, Patel AV, Bush WS, Aldrich MC, Cussenot O, Petrovics G, Cullen J, Neslund-Dudas CM, Stern MC, Kote-Jarai Z, Govindasami K, Cook MB, Chokkalingam AP, Hsing AW, Goodman PJ, Hoffmann TJ, Drake BF, Hu JJ, Keaton JM, Hellwege JN, Clark PE, Jalloh M, Gueye SM, Niang L, Ogunbiyi O, Idowu MO, Popoola O, Adebiyi AO, Aisuodionoe-Shadrach OI, Ajibola HO, Jamda MA, Oluwole OP, Nwegbu M, Adusei B, Mante S, Darkwa-Abrahams A, Mensah JE, Diop H, Van Den Eeden SK, Blanchet P, Fowke JH, Casey G, Hennis AJ, Lubwama A, Thompson IM Jr, Leach R, Easton DF, Preuss MH, Loos RJ, Gundell SM, Wan P, Mohler JL, Fontham ET, Smith GJ, Taylor JA, Srivastava S, Eeles RA, Carpten JD, Kibel AS, Multigner L, Parent ME, Menegaux F, Cancel-Tassin G, Klein EA, Andrews C, Rebbeck TR, Brureau L, Ambs S, Edwards TL, Watya S, Chanock SJ, Witte JS, Blot WJ, Michael Gaziano J, Justice AC, Conti DV, Haiman CA. Evidence of Novel Susceptibility Variants for Prostate Cancer and a Multiancestry Polygenic Risk Score Associated with Aggressive Disease in Men of African Ancestry. Eur Urol. 2023 Jul;84(1):13-21. doi: 10.1016/j.eururo.2023.01.022. Epub 2023 Mar 3. PMID 36872133
- [Background] Fang S, Yarmolinsky J, Gill D, Bull CJ, Perks CM; PRACTICAL Consortium; Davey Smith G, Gaunt TR, Richardson TG. Association between genetically proxied PCSK9 inhibition and prostate cancer risk: A Mendelian randomisation study. PLoS Med. 2023 Jan 3;20(1):e1003988. doi: 10.1371/journal.pmed.1003988. eCollection 2023 Jan. PMID 36595504
- [Background] Abdi B, Basset N, Perrot E, Benderra MA, Khalil A, Oudard S, Blanchet P, Brureau L, Coulet F, Cussenot O, Cancel-Tassin G. DNA damage repair gene germline profiling for metastatic prostate cancer patients of different ancestries. Prostate. 2022 Sep;82(12):1196-1201. doi: 10.1002/pros.24374. Epub 2022 Jun 2. PMID 35652560
- [Background] Burns D, Anokian E, Saunders EJ, Bristow RG, Fraser M, Reimand J, Schlomm T, Sauter G, Brors B, Korbel J, Weischenfeldt J, Waszak SM, Corcoran NM, Jung CH, Pope BJ, Hovens CM, Cancel-Tassin G, Cussenot O, Loda M, Sander C, Hayes VM, Dalsgaard Sorensen K, Lu YJ, Hamdy FC, Foster CS, Gnanapragasam V, Butler A, Lynch AG, Massie CE; CR-UK/Prostate Cancer UK, ICGC, The PPCG; Woodcock DJ, Cooper CS, Wedge DC, Brewer DS, Kote-Jarai Z, Eeles RA. Rare Germline Variants Are Associated with Rapid Biochemical Recurrence After Radical Prostate Cancer Treatment: A Pan Prostate Cancer Group Study. Eur Urol. 2022 Aug;82(2):201-211. doi: 10.1016/j.eururo.2022.05.007. Epub 2022 May 31. PMID 35659150
- [Background] Kuhl V, Clegg W, Meek S, Lenz L, Flake DD 2nd, Ronan T, Kornilov M, Horsch D, Scheer M, Farber D, Zalaznick H, Cussenot O, Comperat E, Cancel-Tassin G, Wild PJ, Chun FK, Mandel P, Moinfar F, Cohen T, Delee S, Kronenwett R, Doedt J. Development and validation of a cell cycle progression signature for decentralized testing of men with prostate cancer. Biomark Med. 2022 Apr;16(6):449-459. doi: 10.2217/bmm-2021-0479. Epub 2022 Mar 24. PMID 35321552
- [Background] Huynh-Le MP, Karunamuni R, Fan CC, Asona L, Thompson WK, Martinez ME, Eeles RA, Kote-Jarai Z, Muir KR, Lophatananon A, Schleutker J, Pashayan N, Batra J, Gronberg H, Neal DE, Nordestgaard BG, Tangen CM, MacInnis RJ, Wolk A, Albanes D, Haiman CA, Travis RC, Blot WJ, Stanford JL, Mucci LA, West CML, Nielsen SF, Kibel AS, Cussenot O, Berndt SI, Koutros S, Sorensen KD, Cybulski C, Grindedal EM, Menegaux F, Park JY, Ingles SA, Maier C, Hamilton RJ, Rosenstein BS, Lu YJ, Watya S, Vega A, Kogevinas M, Wiklund F, Penney KL, Huff CD, Teixeira MR, Multigner L, Leach RJ, Brenner H, John EM, Kaneva R, Logothetis CJ, Neuhausen SL, De Ruyck K, Ost P, Razack A, Newcomb LF, Fowke JH, Gamulin M, Abraham A, Claessens F, Castelao JE, Townsend PA, Crawford DC, Petrovics G, van Schaik RHN, Parent ME, Hu JJ, Zheng W; UKGPCS collaborators; APCB (Australian Prostate Cancer BioResource); NC-LA PCaP Investigators; IMPACT Study Steering Committee and Collaborators; Canary PASS Investigators; Profile Study Steering Committee; PRACTICAL Consortium; Mills IG, Andreassen OA, Dale AM, Seibert TM. Prostate cancer risk stratification improvement across multiple ancestries with new polygenic hazard score. Prostate Cancer Prostatic Dis. 2022 Apr;25(4):755-761. doi: 10.1038/s41391-022-00497-7. Epub 2022 Feb 12. PMID 35152271
- [Background] Karunamuni RA, Huynh-Le MP, Fan CC, Thompson W, Lui A, Martinez ME, Rose BS, Mahal B, Eeles RA, Kote-Jarai Z, Muir K, Lophatananon A; UKGPCS Collaborators; Tangen CM, Goodman PJ, Thompson IM Jr, Blot WJ, Zheng W, Kibel AS, Drake BF, Cussenot O, Cancel-Tassin G, Menegaux F, Truong T, Park JY, Lin HY, Taylor JA, Bensen JT, Mohler JL, Fontham ETH, Multigner L, Blanchet P, Brureau L, Romana M, Leach RJ, John EM, Fowke JH, Bush WS, Aldrich MC, Crawford DC, Cullen J, Petrovics G, Parent ME, Hu JJ, Sanderson M; PRACTICAL Consortium; Mills IG, Andreassen OA, Dale AM, Seibert TM. Performance of African-ancestry-specific polygenic hazard score varies according to local ancestry in 8q24. Prostate Cancer Prostatic Dis. 2022 Feb;25(2):229-237. doi: 10.1038/s41391-021-00403-7. Epub 2021 Jun 14. PMID 34127801
- [Background] Darst BF, Hughley R, Pfennig A, Hazra U, Fan C, Wan P, Sheng X, Xia L, Andrews C, Chen F, Berndt SI, Kote-Jarai Z, Govindasami K, Bensen JT, Ingles SA, Rybicki BA, Nemesure B, John EM, Fowke JH, Huff CD, Strom SS, Isaacs WB, Park JY, Zheng W, Ostrander EA, Walsh PC, Carpten J, Sellers TA, Yamoah K, Murphy AB, Sanderson M, Crawford DC, Gapstur SM, Bush WS, Aldrich MC, Cussenot O, Petrovics G, Cullen J, Neslund-Dudas C, Kittles RA, Xu J, Stern MC, Chokkalingam AP, Multigner L, Parent ME, Menegaux F, Cancel-Tassin G, Kibel AS, Klein EA, Goodman PJ, Stanford JL, Drake BF, Hu JJ, Clark PE, Blanchet P, Casey G, Hennis AJM, Lubwama A, Thompson IM Jr, Leach RJ, Gundell SM, Pooler L, Mohler JL, Fontham ETH, Smith GJ, Taylor JA, Brureau L, Blot WJ, Biritwum R, Tay E, Truelove A, Niwa S, Tettey Y, Varma R, McKean-Cowdin R, Torres M, Jalloh M, Magueye Gueye S, Niang L, Ogunbiyi O, Oladimeji Idowu M, Popoola O, Adebiyi AO, Aisuodionoe-Shadrach OI, Nwegbu M, Adusei B, Mante S, Darkwa-Abrahams A, Yeboah ED, Mensah JE, Anthony Adjei A, Diop H, Cook MB, Chanock SJ, Watya S, Eeles RA, Chiang CWK, Lachance J, Rebbeck TR, Conti DV, Haiman CA. A Rare Germline HOXB13 Variant Contributes to Risk of Prostate Cancer in Men of African Ancestry. Eur Urol. 2022 May;81(5):458-462. doi: 10.1016/j.eururo.2021.12.023. Epub 2022 Jan 12. PMID 35031163
- [Background] Karlsson Q, Brook MN, Dadaev T, Wakerell S, Saunders EJ, Muir K, Neal DE, Giles GG, MacInnis RJ, Thibodeau SN, McDonnell SK, Cannon-Albright L, Teixeira MR, Paulo P, Cardoso M, Huff C, Li D, Yao Y, Scheet P, Permuth JB, Stanford JL, Dai JY, Ostrander EA, Cussenot O, Cancel-Tassin G, Hoegel J, Herkommer K, Schleutker J, Tammela TLJ, Rathinakannan V, Sipeky C, Wiklund F, Gronberg H, Aly M, Isaacs WB, Dickinson JL, FitzGerald LM, Chua MLK, Nguyen-Dumont T; PRACTICAL Consortium; Schaid DJ, Southey MC, Eeles RA, Kote-Jarai Z. Rare Germline Variants in ATM Predispose to Prostate Cancer: A PRACTICAL Consortium Study. Eur Urol Oncol. 2021 Aug;4(4):570-579. doi: 10.1016/j.euo.2020.12.001. Epub 2021 Jan 9. PMID 33436325
- [Background] Wang V, Geybels MS, Jordahl KM, Gerke T, Hamid A, Penney KL, Markt SC, Freedman M, Pomerantz M, Lee GM, Rana H, Bornigen D, Rebbeck TR, Huttenhower C, Eeles RA, Stanford JL, Consortium P, Berndt SI, Claessens F, Sorensen KD, Park JY, Vega A, Usmani N, Mucci L, Sweeney CJ. A polymorphism in the promoter of FRAS1 is a candidate SNP associated with metastatic prostate cancer. Prostate. 2021 Jul;81(10):683-693. doi: 10.1002/pros.24148. Epub 2021 May 6. PMID 33956343
- [Background] Karunamuni RA, Huynh-Le MP, Fan CC, Thompson W, Eeles RA, Kote-Jarai Z, Muir K, Lophatananon A; UKGPCS collaborators; Schleutker J, Pashayan N, Batra J; APCB BioResource (Australian Prostate Cancer BioResource); Gronberg H, Walsh EI, Turner EL, Lane A, Martin RM, Neal DE, Donovan JL, Hamdy FC, Nordestgaard BG, Tangen CM, MacInnis RJ, Wolk A, Albanes D, Haiman CA, Travis RC, Stanford JL, Mucci LA, West CML, Nielsen SF, Kibel AS, Wiklund F, Cussenot O, Berndt SI, Koutros S, Sorensen KD, Cybulski C, Grindedal EM, Park JY, Ingles SA, Maier C, Hamilton RJ, Rosenstein BS, Vega A; IMPACT Study Steering Committee and Collaborators; Kogevinas M, Penney KL, Teixeira MR, Brenner H, John EM, Kaneva R, Logothetis CJ, Neuhausen SL, Razack A, Newcomb LF; Canary PASS Investigators; Gamulin M, Usmani N, Claessens F, Gago-Dominguez M, Townsend PA, Roobol MJ, Zheng W; Profile Study Steering Committee; Mills IG, Andreassen OA, Dale AM, Seibert TM; PRACTICAL Consortium. Additional SNPs improve risk stratification of a polygenic hazard score for prostate cancer. Prostate Cancer Prostatic Dis. 2021 Jun;24(2):532-541. doi: 10.1038/s41391-020-00311-2. Epub 2021 Jan 8. PMID 33420416
- [Background] Lotan TL, Kaur HB, Salles DC, Murali S, Schaeffer EM, Lanchbury JS, Isaacs WB, Brown R, Richardson AL, Cussenot O, Cancel-Tassin G, Timms KM, Antonarakis ES. Homologous recombination deficiency (HRD) score in germline BRCA2- versus ATM-altered prostate cancer. Mod Pathol. 2021 Jun;34(6):1185-1193. doi: 10.1038/s41379-020-00731-4. Epub 2021 Jan 18. PMID 33462368
- [Background] Leon P, Cancel-Tassin G, Bourdon V, Buecher B, Oudard S, Brureau L, Jouffe L, Blanchet P, Stoppa-Lyonnet D, Coulet F, Sobol H, Cussenot O. Bayesian predictive model to assess BRCA2 mutational status according to clinical history: Early onset, metastatic phenotype or family history of breast/ovary cancer. Prostate. 2021 May;81(6):318-325. doi: 10.1002/pros.24109. Epub 2021 Feb 18. PMID 33599307
- [Background] Schaid DJ, McDonnell SK, FitzGerald LM, DeRycke L, Fogarty Z, Giles GG, MacInnis RJ, Southey MC, Nguyen-Dumont T, Cancel-Tassin G, Cussenot O, Whittemore AS, Sieh W, Ioannidis NM, Hsieh CL, Stanford JL, Schleutker J, Cropp CD, Carpten J, Hoegel J, Eeles R, Kote-Jarai Z, Ackerman MJ, Klein CJ, Mandal D, Cooney KA, Bailey-Wilson JE, Helfand B, Catalona WJ, Wiklund F, Riska S, Bahetti S, Larson MC, Cannon Albright L, Teerlink C, Xu J, Isaacs W, Ostrander EA, Thibodeau SN. Two-stage Study of Familial Prostate Cancer by Whole-exome Sequencing and Custom Capture Identifies 10 Novel Genes Associated with the Risk of Prostate Cancer. Eur Urol. 2021 Mar;79(3):353-361. doi: 10.1016/j.eururo.2020.07.038. Epub 2020 Aug 14. PMID 32800727
- [Background] Conti DV, Darst BF, Moss LC, Saunders EJ, Sheng X, Chou A, Schumacher FR, Olama AAA, Benlloch S, Dadaev T, Brook MN, Sahimi A, Hoffmann TJ, Takahashi A, Matsuda K, Momozawa Y, Fujita M, Muir K, Lophatananon A, Wan P, Le Marchand L, Wilkens LR, Stevens VL, Gapstur SM, Carter BD, Schleutker J, Tammela TLJ, Sipeky C, Auvinen A, Giles GG, Southey MC, MacInnis RJ, Cybulski C, Wokolorczyk D, Lubinski J, Neal DE, Donovan JL, Hamdy FC, Martin RM, Nordestgaard BG, Nielsen SF, Weischer M, Bojesen SE, Roder MA, Iversen P, Batra J, Chambers S, Moya L, Horvath L, Clements JA, Tilley W, Risbridger GP, Gronberg H, Aly M, Szulkin R, Eklund M, Nordstrom T, Pashayan N, Dunning AM, Ghoussaini M, Travis RC, Key TJ, Riboli E, Park JY, Sellers TA, Lin HY, Albanes D, Weinstein SJ, Mucci LA, Giovannucci E, Lindstrom S, Kraft P, Hunter DJ, Penney KL, Turman C, Tangen CM, Goodman PJ, Thompson IM Jr, Hamilton RJ, Fleshner NE, Finelli A, Parent ME, Stanford JL, Ostrander EA, Geybels MS, Koutros S, Freeman LEB, Stampfer M, Wolk A, Hakansson N, Andriole GL, Hoover RN, Machiela MJ, Sorensen KD, Borre M, Blot WJ, Zheng W, Yeboah ED, Mensah JE, Lu YJ, Zhang HW, Feng N, Mao X, Wu Y, Zhao SC, Sun Z, Thibodeau SN, McDonnell SK, Schaid DJ, West CML, Burnet N, Barnett G, Maier C, Schnoeller T, Luedeke M, Kibel AS, Drake BF, Cussenot O, Cancel-Tassin G, Menegaux F, Truong T, Koudou YA, John EM, Grindedal EM, Maehle L, Khaw KT, Ingles SA, Stern MC, Vega A, Gomez-Caamano A, Fachal L, Rosenstein BS, Kerns SL, Ostrer H, Teixeira MR, Paulo P, Brandao A, Watya S, Lubwama A, Bensen JT, Fontham ETH, Mohler J, Taylor JA, Kogevinas M, Llorca J, Castano-Vinyals G, Cannon-Albright L, Teerlink CC, Huff CD, Strom SS, Multigner L, Blanchet P, Brureau L, Kaneva R, Slavov C, Mitev V, Leach RJ, Weaver B, Brenner H, Cuk K, Holleczek B, Saum KU, Klein EA, Hsing AW, Kittles RA, Murphy AB, Logothetis CJ, Kim J, Neuhausen SL, Steele L, Ding YC, Isaacs WB, Nemesure B, Hennis AJM, Carpten J, Pandha H, Michael A, De Ruyck K, De Meerleer G, Ost P, Xu J, Razack A, Lim J, Teo SH, Newcomb LF, Lin DW, Fowke JH, Neslund-Dudas C, Rybicki BA, Gamulin M, Lessel D, Kulis T, Usmani N, Singhal S, Parliament M, Claessens F, Joniau S, Van den Broeck T, Gago-Dominguez M, Castelao JE, Martinez ME, Larkin S, Townsend PA, Aukim-Hastie C, Bush WS, Aldrich MC, Crawford DC, Srivastava S, Cullen JC, Petrovics G, Casey G, Roobol MJ, Jenster G, van Schaik RHN, Hu JJ, Sanderson M, Varma R, McKean-Cowdin R, Torres M, Mancuso N, Berndt SI, Van Den Eeden SK, Easton DF, Chanock SJ, Cook MB, Wiklund F, Nakagawa H, Witte JS, Eeles RA, Kote-Jarai Z, Haiman CA. Trans-ancestry genome-wide association meta-analysis of prostate cancer identifies new susceptibility loci and informs genetic risk prediction. Nat Genet. 2021 Jan;53(1):65-75. doi: 10.1038/s41588-020-00748-0. Epub 2021 Jan 4. PMID 33398198
- [Background] Karunamuni RA, Huynh-Le MP, Fan CC, Thompson W, Eeles RA, Kote-Jarai Z, Muir K; UKGPCS Collaborators; Lophatananon A, Tangen CM, Goodman PJ, Thompson IM Jr, Blot WJ, Zheng W, Kibel AS, Drake BF, Cussenot O, Cancel-Tassin G, Menegaux F, Truong T, Park JY, Lin HY, Bensen JT, Fontham ETH, Mohler JL, Taylor JA, Multigner L, Blanchet P, Brureau L, Romana M, Leach RJ, John EM, Fowke J, Bush WS, Aldrich M, Crawford DC, Srivastava S, Cullen JC, Petrovics G, Parent ME, Hu JJ, Sanderson M, Mills IG, Andreassen OA, Dale AM, Seibert TM; PRACTICAL Consortium. African-specific improvement of a polygenic hazard score for age at diagnosis of prostate cancer. Int J Cancer. 2021 Jan 1;148(1):99-105. doi: 10.1002/ijc.33282. Epub 2020 Sep 24. PMID 32930425
- [Background] Brandao A, Paulo P, Maia S, Pinheiro M, Peixoto A, Cardoso M, Silva MP, Santos C, Eeles RA, Kote-Jarai Z, Muir K, Ukgpcs Collaborators, Schleutker J, Wang Y, Pashayan N, Batra J, Apcb BioResource, Gronberg H, Neal DE, Nordestgaard BG, Tangen CM, Southey MC, Wolk A, Albanes D, Haiman CA, Travis RC, Stanford JL, Mucci LA, West CML, Nielsen SF, Kibel AS, Cussenot O, Berndt SI, Koutros S, Sorensen KD, Cybulski C, Grindedal EM, Park JY, Ingles SA, Maier C, Hamilton RJ, Rosenstein BS, Vega A, The Impact Study Steering Committee And Collaborators, Kogevinas M, Wiklund F, Penney KL, Brenner H, John EM, Kaneva R, Logothetis CJ, Neuhausen SL, Ruyck K, Razack A, Newcomb LF, Canary Pass Investigators, Lessel D, Usmani N, Claessens F, Gago-Dominguez M, Townsend PA, Roobol MJ, The Profile Study Steering Committee, The Practical Consortium, Teixeira MR. The CHEK2 Variant C.349A>G Is Associated with Prostate Cancer Risk and Carriers Share a Common Ancestor. Cancers (Basel). 2020 Nov 4;12(11):3254. doi: 10.3390/cancers12113254. PMID 33158149
- [Background] Darst BF, Wan P, Sheng X, Bensen JT, Ingles SA, Rybicki BA, Nemesure B, John EM, Fowke JH, Stevens VL, Berndt SI, Huff CD, Strom SS, Park JY, Zheng W, Ostrander EA, Walsh PC, Srivastava S, Carpten J, Sellers TA, Yamoah K, Murphy AB, Sanderson M, Crawford DC, Gapstur SM, Bush WS, Aldrich MC, Cussenot O, Yeager M, Petrovics G, Cullen J, Neslund-Dudas C, Kittles RA, Xu J, Stern MC, Kote-Jarai Z, Govindasami K, Chokkalingam AP, Multigner L, Parent ME, Menegaux F, Cancel-Tassin G, Kibel AS, Klein EA, Goodman PJ, Drake BF, Hu JJ, Clark PE, Blanchet P, Casey G, Hennis AJM, Lubwama A, Thompson IM Jr, Leach R, Gundell SM, Pooler L, Xia L, Mohler JL, Fontham ETH, Smith GJ, Taylor JA, Eeles RA, Brureau L, Chanock SJ, Watya S, Stanford JL, Mandal D, Isaacs WB, Cooney K, Blot WJ, Conti DV, Haiman CA. A Germline Variant at 8q24 Contributes to Familial Clustering of Prostate Cancer in Men of African Ancestry. Eur Urol. 2020 Sep;78(3):316-320. doi: 10.1016/j.eururo.2020.04.060. Epub 2020 May 12. PMID 32409115
- [Background] Wu L, Yang Y, Guo X, Shu XO, Cai Q, Shu X, Li B, Tao R, Wu C, Nikas JB, Sun Y, Zhu J, Roobol MJ, Giles GG, Brenner H, John EM, Clements J, Grindedal EM, Park JY, Stanford JL, Kote-Jarai Z, Haiman CA, Eeles RA, Zheng W, Long J; PRACTICAL consortium; CRUK Consortium; BPC3 Consortium; CAPS Consortium; PEGASUS Consortium. An integrative multi-omics analysis to identify candidate DNA methylation biomarkers related to prostate cancer risk. Nat Commun. 2020 Aug 6;11(1):3905. doi: 10.1038/s41467-020-17673-9. PMID 32764609
- [Background] Ahmed M, Goh C, Saunders E, Cieza-Borrella C; PRACTICAL consortium; Kote-Jarai Z, Schumacher FR, Eeles R. Germline genetic variation in prostate susceptibility does not predict outcomes in the chemoprevention trials PCPT and SELECT. Prostate Cancer Prostatic Dis. 2020 Jun;23(2):333-342. doi: 10.1038/s41391-019-0181-y. Epub 2019 Nov 27. PMID 31776447
- [Background] Wu L, Wang J, Cai Q, Cavazos TB, Emami NC, Long J, Shu XO, Lu Y, Guo X, Bauer JA, Pasaniuc B, Penney KL, Freedman ML, Kote-Jarai Z, Witte JS, Haiman CA, Eeles RA, Zheng W; PRACTICAL, CRUK, BPC3, CAPS, PEGASUS Consortia. Identification of Novel Susceptibility Loci and Genes for Prostate Cancer Risk: A Transcriptome-Wide Association Study in Over 140,000 European Descendants. Cancer Res. 2019 Jul 1;79(13):3192-3204. doi: 10.1158/0008-5472.CAN-18-3536. Epub 2019 May 17. PMID 31101764
- [Background] Matejcic M, Saunders EJ, Dadaev T, Brook MN, Wang K, Sheng X, Olama AAA, Schumacher FR, Ingles SA, Govindasami K, Benlloch S, Berndt SI, Albanes D, Koutros S, Muir K, Stevens VL, Gapstur SM, Tangen CM, Batra J, Clements J, Gronberg H, Pashayan N, Schleutker J, Wolk A, West C, Mucci L, Kraft P, Cancel-Tassin G, Sorensen KD, Maehle L, Grindedal EM, Strom SS, Neal DE, Hamdy FC, Donovan JL, Travis RC, Hamilton RJ, Rosenstein B, Lu YJ, Giles GG, Kibel AS, Vega A, Bensen JT, Kogevinas M, Penney KL, Park JY, Stanford JL, Cybulski C, Nordestgaard BG, Brenner H, Maier C, Kim J, Teixeira MR, Neuhausen SL, De Ruyck K, Razack A, Newcomb LF, Lessel D, Kaneva R, Usmani N, Claessens F, Townsend PA, Gago-Dominguez M, Roobol MJ, Menegaux F, Khaw KT, Cannon-Albright LA, Pandha H, Thibodeau SN, Schaid DJ; PRACTICAL (Prostate Cancer Association Group to Investigate Cancer-Associated Alterations in the Genome) Consortium; Wiklund F, Chanock SJ, Easton DF, Eeles RA, Kote-Jarai Z, Conti DV, Haiman CA. Germline variation at 8q24 and prostate cancer risk in men of European ancestry. Nat Commun. 2018 Nov 5;9(1):4616. doi: 10.1038/s41467-018-06863-1. PMID 30397198
- [Background] Kamoun A, Cancel-Tassin G, Fromont G, Elarouci N, Armenoult L, Ayadi M, Irani J, Leroy X, Villers A, Fournier G, Doucet L, Boyault S, Brureau L, Multigner L, Diedhiou A, Roupret M, Comperat E, Blanchet P, de Reynies A, Cussenot O. Comprehensive molecular classification of localized prostate adenocarcinoma reveals a tumour subtype predictive of non-aggressive disease. Ann Oncol. 2018 Aug 1;29(8):1814-1821. doi: 10.1093/annonc/mdy224. PMID 29945238
- [Background] Schumacher FR, Al Olama AA, Berndt SI, Benlloch S, Ahmed M, Saunders EJ, Dadaev T, Leongamornlert D, Anokian E, Cieza-Borrella C, Goh C, Brook MN, Sheng X, Fachal L, Dennis J, Tyrer J, Muir K, Lophatananon A, Stevens VL, Gapstur SM, Carter BD, Tangen CM, Goodman PJ, Thompson IM Jr, Batra J, Chambers S, Moya L, Clements J, Horvath L, Tilley W, Risbridger GP, Gronberg H, Aly M, Nordstrom T, Pharoah P, Pashayan N, Schleutker J, Tammela TLJ, Sipeky C, Auvinen A, Albanes D, Weinstein S, Wolk A, Hakansson N, West CML, Dunning AM, Burnet N, Mucci LA, Giovannucci E, Andriole GL, Cussenot O, Cancel-Tassin G, Koutros S, Beane Freeman LE, Sorensen KD, Orntoft TF, Borre M, Maehle L, Grindedal EM, Neal DE, Donovan JL, Hamdy FC, Martin RM, Travis RC, Key TJ, Hamilton RJ, Fleshner NE, Finelli A, Ingles SA, Stern MC, Rosenstein BS, Kerns SL, Ostrer H, Lu YJ, Zhang HW, Feng N, Mao X, Guo X, Wang G, Sun Z, Giles GG, Southey MC, MacInnis RJ, FitzGerald LM, Kibel AS, Drake BF, Vega A, Gomez-Caamano A, Szulkin R, Eklund M, Kogevinas M, Llorca J, Castano-Vinyals G, Penney KL, Stampfer M, Park JY, Sellers TA, Lin HY, Stanford JL, Cybulski C, Wokolorczyk D, Lubinski J, Ostrander EA, Geybels MS, Nordestgaard BG, Nielsen SF, Weischer M, Bisbjerg R, Roder MA, Iversen P, Brenner H, Cuk K, Holleczek B, Maier C, Luedeke M, Schnoeller T, Kim J, Logothetis CJ, John EM, Teixeira MR, Paulo P, Cardoso M, Neuhausen SL, Steele L, Ding YC, De Ruyck K, De Meerleer G, Ost P, Razack A, Lim J, Teo SH, Lin DW, Newcomb LF, Lessel D, Gamulin M, Kulis T, Kaneva R, Usmani N, Singhal S, Slavov C, Mitev V, Parliament M, Claessens F, Joniau S, Van den Broeck T, Larkin S, Townsend PA, Aukim-Hastie C, Gago-Dominguez M, Castelao JE, Martinez ME, Roobol MJ, Jenster G, van Schaik RHN, Menegaux F, Truong T, Koudou YA, Xu J, Khaw KT, Cannon-Albright L, Pandha H, Michael A, Thibodeau SN, McDonnell SK, Schaid DJ, Lindstrom S, Turman C, Ma J, Hunter DJ, Riboli E, Siddiq A, Canzian F, Kolonel LN, Le Marchand L, Hoover RN, Machiela MJ, Cui Z, Kraft P, Amos CI, Conti DV, Easton DF, Wiklund F, Chanock SJ, Henderson BE, Kote-Jarai Z, Haiman CA, Eeles RA; Profile Study; Australian Prostate Cancer BioResource (APCB); IMPACT Study; Canary PASS Investigators; Breast and Prostate Cancer Cohort Consortium (BPC3); PRACTICAL (Prostate Cancer Association Group to Investigate Cancer-Associated Alterations in the Genome) Consortium; Cancer of the Prostate in Sweden (CAPS); Prostate Cancer Genome-wide Association Study of Uncommon Susceptibility Loci (PEGASUS); Genetic Associations and Mechanisms in Oncology (GAME-ON)/Elucidating Loci Involved in Prostate Cancer Susceptibility (ELLIPSE) Consortium. Association analyses of more than 140,000 men identify 63 new prostate cancer susceptibility loci. Nat Genet. 2018 Jul;50(7):928-936. doi: 10.1038/s41588-018-0142-8. Epub 2018 Jun 11. PMID 29892016
- [Background] Dadaev T, Saunders EJ, Newcombe PJ, Anokian E, Leongamornlert DA, Brook MN, Cieza-Borrella C, Mijuskovic M, Wakerell S, Olama AAA, Schumacher FR, Berndt SI, Benlloch S, Ahmed M, Goh C, Sheng X, Zhang Z, Muir K, Govindasami K, Lophatananon A, Stevens VL, Gapstur SM, Carter BD, Tangen CM, Goodman P, Thompson IM Jr, Batra J, Chambers S, Moya L, Clements J, Horvath L, Tilley W, Risbridger G, Gronberg H, Aly M, Nordstrom T, Pharoah P, Pashayan N, Schleutker J, Tammela TLJ, Sipeky C, Auvinen A, Albanes D, Weinstein S, Wolk A, Hakansson N, West C, Dunning AM, Burnet N, Mucci L, Giovannucci E, Andriole G, Cussenot O, Cancel-Tassin G, Koutros S, Freeman LEB, Sorensen KD, Orntoft TF, Borre M, Maehle L, Grindedal EM, Neal DE, Donovan JL, Hamdy FC, Martin RM, Travis RC, Key TJ, Hamilton RJ, Fleshner NE, Finelli A, Ingles SA, Stern MC, Rosenstein B, Kerns S, Ostrer H, Lu YJ, Zhang HW, Feng N, Mao X, Guo X, Wang G, Sun Z, Giles GG, Southey MC, MacInnis RJ, FitzGerald LM, Kibel AS, Drake BF, Vega A, Gomez-Caamano A, Fachal L, Szulkin R, Eklund M, Kogevinas M, Llorca J, Castano-Vinyals G, Penney KL, Stampfer M, Park JY, Sellers TA, Lin HY, Stanford JL, Cybulski C, Wokolorczyk D, Lubinski J, Ostrander EA, Geybels MS, Nordestgaard BG, Nielsen SF, Weisher M, Bisbjerg R, Roder MA, Iversen P, Brenner H, Cuk K, Holleczek B, Maier C, Luedeke M, Schnoeller T, Kim J, Logothetis CJ, John EM, Teixeira MR, Paulo P, Cardoso M, Neuhausen SL, Steele L, Ding YC, De Ruyck K, De Meerleer G, Ost P, Razack A, Lim J, Teo SH, Lin DW, Newcomb LF, Lessel D, Gamulin M, Kulis T, Kaneva R, Usmani N, Slavov C, Mitev V, Parliament M, Singhal S, Claessens F, Joniau S, Van den Broeck T, Larkin S, Townsend PA, Aukim-Hastie C, Gago-Dominguez M, Castelao JE, Martinez ME, Roobol MJ, Jenster G, van Schaik RHN, Menegaux F, Truong T, Koudou YA, Xu J, Khaw KT, Cannon-Albright L, Pandha H, Michael A, Kierzek A, Thibodeau SN, McDonnell SK, Schaid DJ, Lindstrom S, Turman C, Ma J, Hunter DJ, Riboli E, Siddiq A, Canzian F, Kolonel LN, Le Marchand L, Hoover RN, Machiela MJ, Kraft P; PRACTICAL (Prostate Cancer Association Group to Investigate Cancer-Associated Alterations in the Genome) Consortium; Freedman M, Wiklund F, Chanock S, Henderson BE, Easton DF, Haiman CA, Eeles RA, Conti DV, Kote-Jarai Z. Fine-mapping of prostate cancer susceptibility loci in a large meta-analysis identifies candidate causal variants. Nat Commun. 2018 Jun 11;9(1):2256. doi: 10.1038/s41467-018-04109-8. PMID 29892050
- [Background] Conti DV, Wang K, Sheng X, Bensen JT, Hazelett DJ, Cook MB, Ingles SA, Kittles RA, Strom SS, Rybicki BA, Nemesure B, Isaacs WB, Stanford JL, Zheng W, Sanderson M, John EM, Park JY, Xu J, Stevens VL, Berndt SI, Huff CD, Wang Z, Yeboah ED, Tettey Y, Biritwum RB, Adjei AA, Tay E, Truelove A, Niwa S, Sellers TA, Yamoah K, Murphy AB, Crawford DC, Gapstur SM, Bush WS, Aldrich MC, Cussenot O, Petrovics G, Cullen J, Neslund-Dudas C, Stern MC, Jarai ZK, Govindasami K, Chokkalingam AP, Hsing AW, Goodman PJ, Hoffmann T, Drake BF, Hu JJ, Clark PE, Van Den Eeden SK, Blanchet P, Fowke JH, Casey G, Hennis AJM, Han Y, Lubwama A, Thompson IM Jr, Leach R, Easton DF, Schumacher F, Van den Berg DJ, Gundell SM, Stram A, Wan P, Xia L, Pooler LC, Mohler JL, Fontham ETH, Smith GJ, Taylor JA, Srivastava S, Eeles RA, Carpten J, Kibel AS, Multigner L, Parent ME, Menegaux F, Cancel-Tassin G, Klein EA, Brureau L, Stram DO, Watya S, Chanock SJ, Witte JS, Blot WJ, Henderson BE, Haiman CA; PRACTICAL/ELLIPSE Consortium. Two Novel Susceptibility Loci for Prostate Cancer in Men of African Ancestry. J Natl Cancer Inst. 2017 Aug 1;109(8):djx084. doi: 10.1093/jnci/djx084. PMID 29117387
- [Background] Cornu JN, Audet-Walsh E, Drouin S, Bigot P, Valeri A, Fournier G, Azzouzi AR, Roupret M, Cormier L, Chanock S, Guillemette C, Cussenot O, Levesque E, Cancel-Tassin G. Correlation between prostate volume and single nucleotide polymorphisms implicated in the steroid pathway. World J Urol. 2017 Feb;35(2):293-298. doi: 10.1007/s00345-016-1869-4. Epub 2016 Jun 8. PMID 27277477
- [Background] Renard Penna R, Cancel-Tassin G, Comperat E, Mozer P, Leon P, Varinot J, Roupret M, Bitker MO, Lucidarme O, Cussenot O. Apparent diffusion coefficient value is a strong predictor of unsuspected aggressiveness of prostate cancer before radical prostatectomy. World J Urol. 2016 Oct;34(10):1389-95. doi: 10.1007/s00345-016-1789-3. Epub 2016 Feb 22. PMID 26902878
- [Background] Larson NB, McDonnell S, Albright LC, Teerlink C, Stanford J, Ostrander EA, Isaacs WB, Xu J, Cooney KA, Lange E, Schleutker J, Carpten JD, Powell I, Bailey-Wilson J, Cussenot O, Cancel-Tassin G, Giles G, MacInnis R, Maier C, Whittemore AS, Hsieh CL, Wiklund F, Catalona WJ, Foulkes W, Mandal D, Eeles R, Kote-Jarai Z, Ackerman MJ, Olson TM, Klein CJ, Thibodeau SN, Schaid DJ. Post hoc Analysis for Detecting Individual Rare Variant Risk Associations Using Probit Regression Bayesian Variable Selection Methods in Case-Control Sequencing Studies. Genet Epidemiol. 2016 Sep;40(6):461-9. doi: 10.1002/gepi.21983. Epub 2016 Jun 17. PMID 27312771
- [Background] Cornu JN, Cancel-Tassin G, Cox DG, Roupret M, Koutlidis N, Bigot P, Valeri A, Ondet V, Gaffory C, Fournier G, Azzouzi AR, Cormier L, Cussenot O. Impact of Body Mass Index, Age, Prostate Volume, and Genetic Polymorphisms on Prostate-specific Antigen Levels in a Control Population. Eur Urol. 2016 Jul;70(1):6-8. doi: 10.1016/j.eururo.2016.01.027. Epub 2016 Feb 2. PMID 26850968
- [Background] Teerlink CC, Leongamornlert D, Dadaev T, Thomas A, Farnham J, Stephenson RA, Riska S, McDonnell SK, Schaid DJ, Catalona WJ, Zheng SL, Cooney KA, Ray AM, Zuhlke KA, Lange EM, Giles GG, Southey MC, Fitzgerald LM, Rinckleb A, Luedeke M, Maier C, Stanford JL, Ostrander EA, Kaikkonen EM, Sipeky C, Tammela T, Schleutker J, Wiley KE, Isaacs SD, Walsh PC, Isaacs WB, Xu J, Cancel-Tassin G, Cussenot O, Mandal D, Laurie C, Laurie C; PRACTICAL consortium; International Consortium for Prostate Cancer Genetics; Thibodeau SN, Eeles RA, Kote-Jarai Z, Cannon-Albright L. Genome-wide association of familial prostate cancer cases identifies evidence for a rare segregating haplotype at 8q24.21. Hum Genet. 2016 Aug;135(8):923-38. doi: 10.1007/s00439-016-1690-6. Epub 2016 Jun 4. PMID 27262462
- [Background] Helfand BT, Roehl KA, Cooper PR, McGuire BB, Fitzgerald LM, Cancel-Tassin G, Cornu JN, Bauer S, Van Blarigan EL, Chen X, Duggan D, Ostrander EA, Gwo-Shu M, Zhang ZF, Chang SC, Jeong S, Fontham ET, Smith G, Mohler JL, Berndt SI, McDonnell SK, Kittles R, Rybicki BA, Freedman M, Kantoff PW, Pomerantz M, Breyer JP, Smith JR, Rebbeck TR, Mercola D, Isaacs WB, Wiklund F, Cussenot O, Thibodeau SN, Schaid DJ, Cannon-Albright L, Cooney KA, Chanock SJ, Stanford JL, Chan JM, Witte J, Xu J, Bensen JT, Taylor JA, Catalona WJ. Associations of prostate cancer risk variants with disease aggressiveness: results of the NCI-SPORE Genetics Working Group analysis of 18,343 cases. Hum Genet. 2015 Apr;134(4):439-50. doi: 10.1007/s00439-015-1534-9. Epub 2015 Feb 26. PMID 25715684
- [Background] Renard-Penna R, Cancel-Tassin G, Comperat E, Varinot J, Leon P, Roupret M, Mozer P, Vaessen C, Lucidarme O, Bitker MO, Cussenot O. Multiparametric Magnetic Resonance Imaging Predicts Postoperative Pathology but Misses Aggressive Prostate Cancers as Assessed by Cell Cycle Progression Score. J Urol. 2015 Dec;194(6):1617-23. doi: 10.1016/j.juro.2015.06.107. Epub 2015 Aug 10. PMID 26272031
- [Background] Seisen T, Roupret M, Brault D, Leon P, Cancel-Tassin G, Comperat E, Renard-Penna R, Mozer P, Guechot J, Cussenot O. Accuracy of the prostate health index versus the urinary prostate cancer antigen 3 score to predict overall and significant prostate cancer at initial biopsy. Prostate. 2015 Jan;75(1):103-11. doi: 10.1002/pros.22898. Epub 2014 Oct 18. PMID 25327361
- [Background] Berndt SI, Wang Z, Yeager M, Alavanja MC, Albanes D, Amundadottir L, Andriole G, Beane Freeman L, Campa D, Cancel-Tassin G, Canzian F, Cornu JN, Cussenot O, Diver WR, Gapstur SM, Gronberg H, Haiman CA, Henderson B, Hutchinson A, Hunter DJ, Key TJ, Kolb S, Koutros S, Kraft P, Le Marchand L, Lindstrom S, Machiela MJ, Ostrander EA, Riboli E, Schumacher F, Siddiq A, Stanford JL, Stevens VL, Travis RC, Tsilidis KK, Virtamo J, Weinstein S, Wilkund F, Xu J, Lilly Zheng S, Yu K, Wheeler W, Zhang H; African Ancestry Prostate Cancer GWAS Consortium; Sampson J, Black A, Jacobs K, Hoover RN, Tucker M, Chanock SJ. Two susceptibility loci identified for prostate cancer aggressiveness. Nat Commun. 2015 May 5;6:6889. doi: 10.1038/ncomms7889. PMID 25939597
- [Background] Teerlink CC, Thibodeau SN, McDonnell SK, Schaid DJ, Rinckleb A, Maier C, Vogel W, Cancel-Tassin G, Egrot C, Cussenot O, Foulkes WD, Giles GG, Hopper JL, Severi G, Eeles R, Easton D, Kote-Jarai Z, Guy M, Cooney KA, Ray AM, Zuhlke KA, Lange EM, Fitzgerald LM, Stanford JL, Ostrander EA, Wiley KE, Isaacs SD, Walsh PC, Isaacs WB, Wahlfors T, Tammela T, Schleutker J, Wiklund F, Gronberg H, Emanuelsson M, Carpten J, Bailey-Wilson J, Whittemore AS, Oakley-Girvan I, Hsieh CL, Catalona WJ, Zheng SL, Jin G, Lu L, Xu J; International Consortium for Prostate Cancer Genetics; Camp NJ, Cannon-Albright LA. Association analysis of 9,560 prostate cancer cases from the International Consortium of Prostate Cancer Genetics confirms the role of reported prostate cancer associated SNPs for familial disease. Hum Genet. 2014 Mar;133(3):347-56. doi: 10.1007/s00439-013-1384-2. Epub 2013 Oct 26. PMID 24162621
- [Background] Cornu JN, Cancel-Tassin G, Egrot C, Gaffory C, Haab F, Cussenot O. Urine TMPRSS2:ERG fusion transcript integrated with PCA3 score, genotyping, and biological features are correlated to the results of prostatic biopsies in men at risk of prostate cancer. Prostate. 2013 Feb 15;73(3):242-9. doi: 10.1002/pros.22563. Epub 2012 Jul 20. PMID 22821767
- [Background] Xu J, Lange EM, Lu L, Zheng SL, Wang Z, Thibodeau SN, Cannon-Albright LA, Teerlink CC, Camp NJ, Johnson AM, Zuhlke KA, Stanford JL, Ostrander EA, Wiley KE, Isaacs SD, Walsh PC, Maier C, Luedeke M, Vogel W, Schleutker J, Wahlfors T, Tammela T, Schaid D, McDonnell SK, DeRycke MS, Cancel-Tassin G, Cussenot O, Wiklund F, Gronberg H, Eeles R, Easton D, Kote-Jarai Z, Whittemore AS, Hsieh CL, Giles GG, Hopper JL, Severi G, Catalona WJ, Mandal D, Ledet E, Foulkes WD, Hamel N, Mahle L, Moller P, Powell I, Bailey-Wilson JE, Carpten JD, Seminara D, Cooney KA, Isaacs WB; International Consortium for Prostate Cancer Genetics. HOXB13 is a susceptibility gene for prostate cancer: results from the International Consortium for Prostate Cancer Genetics (ICPCG). Hum Genet. 2013 Jan;132(1):5-14. doi: 10.1007/s00439-012-1229-4. Epub 2012 Oct 12. PMID 23064873
- [Background] Bailey-Wilson JE, Childs EJ, Cropp CD, Schaid DJ, Xu J, Camp NJ, Cannon-Albright LA, Farnham JM, George A, Powell I, Carpten JD, Giles GG, Hopper JL, Severi G, English DR, Foulkes WD, Maehle L, Moller P, Eeles R, Easton D, Guy M, Edwards S, Badzioch MD, Whittemore AS, Oakley-Girvan I, Hsieh CL, Dimitrov L, Stanford JL, Karyadi DM, Deutsch K, McIntosh L, Ostrander EA, Wiley KE, Isaacs SD, Walsh PC, Thibodeau SN, McDonnell SK, Hebbring S, Lange EM, Cooney KA, Tammela TL, Schleutker J, Maier C, Bochum S, Hoegel J, Gronberg H, Wiklund F, Emanuelsson M, Cancel-Tassin G, Valeri A, Cussenot O, Isaacs WB; International Consortium for Prostate Cancer Genetics. Analysis of Xq27-28 linkage in the international consortium for prostate cancer genetics (ICPCG) families. BMC Med Genet. 2012 Jun 19;13:46. doi: 10.1186/1471-2350-13-46. PMID 22712434
- [Background] Yates DR, Roupret M, Drouin SJ, Comperat E, Ricci S, Lacave R, Sebe P, Cancel-Tassin G, Bitker MO, Cussenot O. Quantitative RT-PCR analysis of PSA and prostate-specific membrane antigen mRNA to detect circulating tumor cells improves recurrence-free survival nomogram prediction after radical prostatectomy. Prostate. 2012 Sep 1;72(12):1382-8. doi: 10.1002/pros.22488. Epub 2012 Jan 6. PMID 22228175
- [Background] Wang Z, Parikh H, Jia J, Myers T, Yeager M, Jacobs KB, Hutchinson A, Burdett L, Ghosh A, Thun MJ, Gapstur SM, Ryan Diver W, Virtamo J, Albanes D, Cancel-Tassin G, Valeri A, Cussenot O, Offit K, Giovannucci E, Ma J, Stampfer MJ, Michael Gaziano J, Hunter DJ, Dutra-Clarke A, Kirchhoff T, Alavanja M, Freeman LB, Koutros S, Hoover R, Berndt SI, Hayes RB, Agalliu I, Burk RD, Wacholder S, Thomas G, Amundadottir L. Y chromosome haplogroups and prostate cancer in populations of European and Ashkenazi Jewish ancestry. Hum Genet. 2012 Jul;131(7):1173-85. doi: 10.1007/s00439-012-1139-5. Epub 2012 Jan 24. PMID 22271044
- [Background] Jin G, Lu L, Cooney KA, Ray AM, Zuhlke KA, Lange EM, Cannon-Albright LA, Camp NJ, Teerlink CC, Fitzgerald LM, Stanford JL, Wiley KE, Isaacs SD, Walsh PC, Foulkes WD, Giles GG, Hopper JL, Severi G, Eeles R, Easton D, Kote-Jarai Z, Guy M, Rinckleb A, Maier C, Vogel W, Cancel-Tassin G, Egrot C, Cussenot O, Thibodeau SN, McDonnell SK, Schaid DJ, Wiklund F, Gronberg H, Emanuelsson M, Whittemore AS, Oakley-Girvan I, Hsieh CL, Wahlfors T, Tammela T, Schleutker J, Catalona WJ, Zheng SL, Ostrander EA, Isaacs WB, Xu J; International Consortium for Prostate Cancer Genetics. Validation of prostate cancer risk-related loci identified from genome-wide association studies using family-based association analysis: evidence from the International Consortium for Prostate Cancer Genetics (ICPCG). Hum Genet. 2012 Jul;131(7):1095-103. doi: 10.1007/s00439-011-1136-0. Epub 2011 Dec 25. PMID 22198737
- [Background] Lu L, Cancel-Tassin G, Valeri A, Cussenot O, Lange EM, Cooney KA, Farnham JM, Camp NJ, Cannon-Albright LA, Tammela TL, Schleutker J, Hoegel J, Herkommer K, Maier C, Vogel W, Wiklund F, Emanuelsson M, Gronberg H, Wiley KE, Isaacs SD, Walsh PC, Helfand BT, Kan D, Catalona WJ, Stanford JL, FitzGerald LM, Johanneson B, Deutsch K, McIntosh L, Ostrander EA, Thibodeau SN, McDonnell SK, Hebbring S, Schaid DJ, Whittemore AS, Oakley-Girvan I, Hsieh CL, Powell I, Bailey-Wilson JE, Cropp CD, Simpson C, Carpten JD, Seminara D, Zheng SL, Xu J, Giles GG, Severi G, Hopper JL, English DR, Foulkes WD, Maehle L, Moller P, Badzioch MD, Edwards S, Guy M, Eeles R, Easton D, Isaacs WB; International Consortium for Prostate Cancer Genetics. Chromosomes 4 and 8 implicated in a genome wide SNP linkage scan of 762 prostate cancer families collected by the ICPCG. Prostate. 2012 Mar;72(4):410-26. doi: 10.1002/pros.21443. Epub 2011 Jul 11. PMID 21748754
- [Background] Ciampa J, Yeager M, Jacobs K, Thun MJ, Gapstur S, Albanes D, Virtamo J, Weinstein SJ, Giovannucci E, Willett WC, Cancel-Tassin G, Cussenot O, Valeri A, Hunter D, Hoover R, Thomas G, Chanock S, Holmes C, Chatterjee N. Application of a novel score test for genetic association incorporating gene-gene interaction suggests functionality for prostate cancer susceptibility regions. Hum Hered. 2011;72(3):182-93. doi: 10.1159/000331222. Epub 2011 Nov 11. PMID 22086326
- [Background] Berndt SI, Sampson J, Yeager M, Jacobs KB, Wang Z, Hutchinson A, Chung C, Orr N, Wacholder S, Chatterjee N, Yu K, Kraft P, Feigelson HS, Thun MJ, Diver WR, Albanes D, Virtamo J, Weinstein S, Schumacher FR, Cancel-Tassin G, Cussenot O, Valeri A, Andriole GL, Crawford ED, Haiman C, Henderson B, Kolonel L, Le Marchand L, Siddiq A, Riboli E, Travis RC, Kaaks R, Isaacs W, Isaacs S, Wiley KE, Gronberg H, Wiklund F, Stattin P, Xu J, Zheng SL, Sun J, Vatten LJ, Hveem K, Njolstad I, Gerhard DS, Tucker M, Hayes RB, Hoover RN, Fraumeni JF Jr, Hunter DJ, Thomas G, Chanock SJ. Large-scale fine mapping of the HNF1B locus and prostate cancer risk. Hum Mol Genet. 2011 Aug 15;20(16):3322-9. doi: 10.1093/hmg/ddr213. Epub 2011 May 16. PMID 21576123
- [Background] Chung CC, Ciampa J, Yeager M, Jacobs KB, Berndt SI, Hayes RB, Gonzalez-Bosquet J, Kraft P, Wacholder S, Orr N, Yu K, Hutchinson A, Boland J, Chen Q, Feigelson HS, Thun MJ, Diver WR, Albanes D, Virtamo J, Weinstein S, Schumacher FR, Cancel-Tassin G, Cussenot O, Valeri A, Andriole GL, Crawford ED, Haiman CA, Henderson BE, Kolonel L, Le Marchand L, Siddiq A, Riboli E, Key TJ, Kaaks R, Isaacs WB, Isaacs SD, Gronberg H, Wiklund F, Xu J, Vatten LJ, Hveem K, Njolstad I, Gerhard DS, Tucker M, Hoover RN, Fraumeni JF Jr, Hunter DJ, Thomas G, Chatterjee N, Chanock SJ. Fine mapping of a region of chromosome 11q13 reveals multiple independent loci associated with risk of prostate cancer. Hum Mol Genet. 2011 Jul 15;20(14):2869-78. doi: 10.1093/hmg/ddr189. Epub 2011 Apr 29. PMID 21531787
- [Background] Parikh H, Wang Z, Pettigrew KA, Jia J, Daugherty S, Yeager M, Jacobs KB, Hutchinson A, Burdett L, Cullen M, Qi L, Boland J, Collins I, Albert TJ, Vatten LJ, Hveem K, Njolstad I, Cancel-Tassin G, Cussenot O, Valeri A, Virtamo J, Thun MJ, Feigelson HS, Diver WR, Chatterjee N, Thomas G, Albanes D, Chanock SJ, Hunter DJ, Hoover R, Hayes RB, Berndt SI, Sampson J, Amundadottir L. Fine mapping the KLK3 locus on chromosome 19q13.33 associated with prostate cancer susceptibility and PSA levels. Hum Genet. 2011 Jun;129(6):675-85. doi: 10.1007/s00439-011-0953-5. Epub 2011 Feb 15. PMID 21318478
- [Background] Ciampa J, Yeager M, Amundadottir L, Jacobs K, Kraft P, Chung C, Wacholder S, Yu K, Wheeler W, Thun MJ, Divers WR, Gapstur S, Albanes D, Virtamo J, Weinstein S, Giovannucci E, Willett WC, Cancel-Tassin G, Cussenot O, Valeri A, Hunter D, Hoover R, Thomas G, Chanock S, Chatterjee N. Large-scale exploration of gene-gene interactions in prostate cancer using a multistage genome-wide association study. Cancer Res. 2011 May 1;71(9):3287-95. doi: 10.1158/0008-5472.CAN-10-2646. Epub 2011 Mar 3. PMID 21372204
- [Background] Cornu JN, Drouin S, Cancel-Tassin G, Bigot P, Azzouzi AR, Koutlidis N, Cormier L, Gaffory C, Roupret M, Sebe P, Bitker MO, Haab F, Cussenot O. Impact of genotyping on outcome of prostatic biopsies: a multicenter prospective study. Mol Med. 2011 May-Jun;17(5-6):473-7. doi: 10.2119/molmed.2010.00205. Epub 2011 Feb 4. PMID 21308149
- [Background] Cornu JN, Cancel-Tassin G, Ondet V, Girardet C, Cussenot O. Olfactory detection of prostate cancer by dogs sniffing urine: a step forward in early diagnosis. Eur Urol. 2011 Feb;59(2):197-201. doi: 10.1016/j.eururo.2010.10.006. Epub 2010 Oct 15. PMID 20970246
- [Background] Berthon P, Valeri A, Cohen-Akenine A, Drelon E, Paiss T, Wohr G, Latil A, Millasseau P, Mellah I, Cohen N, Blanche H, Bellane-Chantelot C, Demenais F, Teillac P, Le Duc A, de Petriconi R, Hautmann R, Chumakov I, Bachner L, Maitland NJ, Lidereau R, Vogel W, Fournier G, Mangin P, Cussenot O, et al. Predisposing gene for early-onset prostate cancer, localized on chromosome 1q42.2-43. Am J Hum Genet. 1998 Jun;62(6):1416-24. doi: 10.1086/301879. PMID 9585607
- [Background] Correa-Cerro L, Wohr G, Haussler J, Berthon P, Drelon E, Mangin P, Fournier G, Cussenot O, Kraus P, Just W, Paiss T, Cantu JM, Vogel W. (CAG)nCAA and GGN repeats in the human androgen receptor gene are not associated with prostate cancer in a French-German population. Eur J Hum Genet. 1999 Apr;7(3):357-62. doi: 10.1038/sj.ejhg.5200298. PMID 10234512
- [Background] Correa-Cerro L, Berthon P, Haussler J, Bochum S, Drelon E, Mangin P, Fournier G, Paiss T, Cussenot O, Vogel W. Vitamin D receptor polymorphisms as markers in prostate cancer. Hum Genet. 1999 Sep;105(3):281-7. doi: 10.1007/s004390051102. PMID 10987658
- [Background] Valeri A, Fournier G, Morin V, Morin JF, Drelon E, Mangin P, Teillac P, Berthon P, Cussenot O. Early onset and familial predisposition to prostate cancer significantly enhance the probability for breast cancer in first degree relatives. Int J Cancer. 2000 Jun 15;86(6):883-7. doi: 10.1002/(sici)1097-0215(20000615)86:63.0.co;2-f. PMID 10842206
- [Background] Cancel-Tassin G, Latil A, Valeri A, Mangin P, Fournier G, Berthon P, Cussenot O. PCAP is the major known prostate cancer predisposing locus in families from south and west Europe. Eur J Hum Genet. 2001 Feb;9(2):135-42. doi: 10.1038/sj.ejhg.5200592. PMID 11313747
- [Background] Latil AG, Azzouzi R, Cancel GS, Guillaume EC, Cochan-Priollet B, Berthon PL, Cussenot O. Prostate carcinoma risk and allelic variants of genes involved in androgen biosynthesis and metabolism pathways. Cancer. 2001 Sep 1;92(5):1130-7. doi: 10.1002/1097-0142(20010901)92:53.0.co;2-b. PMID 11571725
- [Background] Cormier L, Guillemin F, Valeri A, Fournier G, Cussenot O, Mangin P, Litwin MS. Impact of prostate cancer screening on health-related quality of life in at-risk families. Urology. 2002 Jun;59(6):901-6. doi: 10.1016/s0090-4295(02)01552-2. PMID 12031378
- [Background] Valeri A, Cormier L, Moineau MP, Cancel-Tassin G, Azzouzi R, Doucet L, Baschet F, Cussenot I, L'Her J, Berthon P, Mangin P, Cussenot O, Morin JF, Fournier G. Targeted screening for prostate cancer in high risk families: early onset is a significant risk factor for disease in first degree relatives. J Urol. 2002 Aug;168(2):483-7. doi: 10.1016/s0022-5347(05)64663-0. PMID 12131293
- [Background] Azzouzi AR, Cochand-Priollet B, Mangin P, Fournier G, Berthon P, Latil A, Cussenot O. Impact of constitutional genetic variation in androgen/oestrogen-regulating genes on age-related changes in human prostate. Eur J Endocrinol. 2002 Oct;147(4):479-84. doi: 10.1530/eje.0.1470479. PMID 12370109
- [Background] Cancel-Tassin G, Latil A, Rousseau F, Mangin P, Bottius E, Escary JL, Berthon P, Cussenot O. Association study of polymorphisms in the human estrogen receptor alpha gene and prostate cancer risk. Eur Urol. 2003 Oct;44(4):487-90. doi: 10.1016/s0302-2838(03)00319-1. PMID 14499686
- [Background] Fromont G, Joulin V, Chantrel-Groussard K, Vallancien G, Guillonneau B, Validire P, Latil A, Cussenot O. Allelic losses in localized prostate cancer: association with prognostic factors. J Urol. 2003 Oct;170(4 Pt 1):1394-7. doi: 10.1097/01.ju.0000083329.89215.91. PMID 14501776
- [Background] Latil A, Chene L, Mangin P, Fournier G, Berthon P, Cussenot O. Extensive analysis of the 13q14 region in human prostate tumors: DNA analysis and quantitative expression of genes lying in the interval of deletion. Prostate. 2003 Sep 15;57(1):39-50. doi: 10.1002/pros.10272. PMID 12886522
- [Background] Valeri A, Briollais L, Azzouzi R, Fournier G, Mangin P, Berthon P, Cussenot O, Demenais F. Segregation analysis of prostate cancer in France: evidence for autosomal dominant inheritance and residual brother-brother dependence. Ann Hum Genet. 2003 Mar;67(Pt 2):125-37. doi: 10.1046/j.1469-1809.2003.00022.x. PMID 12675688
- [Background] Roumier X, Azzouzi R, Valeri A, Guillemin F, Fournier G, Cussenot O, Mangin P, Cormier L. Adherence to an annual PSA screening program over 3 years for brothers and sons of men with prostate cancer. Eur Urol. 2004 Mar;45(3):280-5; author reply 285-6. doi: 10.1016/j.eururo.2003.09.022. PMID 15036671
- [Background] Thuret R, Chantrel-Groussard K, Azzouzi AR, Villette JM, Guimard S, Teillac P, Berthon P, Houlgatte A, Latil A, Cussenot O. Clinical relevance of genetic instability in prostatic cells obtained by prostatic massage in early prostate cancer. Br J Cancer. 2005 Jan 31;92(2):236-40. doi: 10.1038/sj.bjc.6602311. PMID 15655554
- [Background] Fromont G, Chene L, Vidaud M, Vallancien G, Mangin P, Fournier G, Validire P, Latil A, Cussenot O. Differential expression of 37 selected genes in hormone-refractory prostate cancer using quantitative taqman real-time RT-PCR. Int J Cancer. 2005 Mar 20;114(2):174-81. doi: 10.1002/ijc.20704. PMID 15543616
- [Background] Roupret M, Fromont G, Bitker MO, Gattegno B, Vallancien G, Cussenot O. Outcome after radical prostatectomy in young men with or without a family history of prostate cancer. Urology. 2006 May;67(5):1028-32. doi: 10.1016/j.urology.2005.11.035. PMID 16698363
- [Background] Azzouzi AR, Stoppa-Lyonnet D, Roupret M, Larre S, Mangin P, Cussenot O. BRCA2 mutation screening is clinically relevant in breast and early prostate cancer families. Int J Urol. 2007 May;14(5):445-6. doi: 10.1111/j.1442-2042.2006.01712.x. PMID 17511731
- [Background] Cussenot O, Azzouzi AR, Nicolaiew N, Mangin P, Cormier L, Fournier G, Valeri A, Cancel-Tassin G. Low-activity V89L variant in SRD5A2 is associated with aggressive prostate cancer risk: an explanation for the adverse effects observed in chemoprevention trials using 5-alpha-reductase inhibitors. Eur Urol. 2007 Oct;52(4):1082-7. doi: 10.1016/j.eururo.2007.04.008. Epub 2007 Apr 13. PMID 17448593
- [Background] Yeager M, Orr N, Hayes RB, Jacobs KB, Kraft P, Wacholder S, Minichiello MJ, Fearnhead P, Yu K, Chatterjee N, Wang Z, Welch R, Staats BJ, Calle EE, Feigelson HS, Thun MJ, Rodriguez C, Albanes D, Virtamo J, Weinstein S, Schumacher FR, Giovannucci E, Willett WC, Cancel-Tassin G, Cussenot O, Valeri A, Andriole GL, Gelmann EP, Tucker M, Gerhard DS, Fraumeni JF Jr, Hoover R, Hunter DJ, Chanock SJ, Thomas G. Genome-wide association study of prostate cancer identifies a second risk locus at 8q24. Nat Genet. 2007 May;39(5):645-9. doi: 10.1038/ng2022. Epub 2007 Apr 1. PMID 17401363
- [Background] Roupret M, Hupertan V, Yates DR, Catto JW, Rehman I, Meuth M, Ricci S, Lacave R, Cancel-Tassin G, de la Taille A, Rozet F, Cathelineau X, Vallancien G, Hamdy FC, Cussenot O. Molecular detection of localized prostate cancer using quantitative methylation-specific PCR on urinary cells obtained following prostate massage. Clin Cancer Res. 2007 Mar 15;13(6):1720-5. doi: 10.1158/1078-0432.CCR-06-2467. PMID 17363525
- [Background] Cussenot O, Azzouzi AR, Bantsimba-Malanda G, Gaffory C, Mangin P, Cormier L, Fournier G, Valeri A, Jouffe L, Roupret M, Fromont G, Sibony M, Comperat E, Cancel-Tassin G. Effect of genetic variability within 8q24 on aggressiveness patterns at diagnosis and familial status of prostate cancer. Clin Cancer Res. 2008 Sep 1;14(17):5635-9. doi: 10.1158/1078-0432.CCR-07-4999. PMID 18765558
- [Background] Ahn J, Berndt SI, Wacholder S, Kraft P, Kibel AS, Yeager M, Albanes D, Giovannucci E, Stampfer MJ, Virtamo J, Thun MJ, Feigelson HS, Cancel-Tassin G, Cussenot O, Thomas G, Hunter DJ, Fraumeni JF Jr, Hoover RN, Chanock SJ, Hayes RB. Variation in KLK genes, prostate-specific antigen and risk of prostate cancer. Nat Genet. 2008 Sep;40(9):1032-4; author reply 1035-6. doi: 10.1038/ng0908-1032. No abstract available. PMID 19165914
- [Background] Fromont G, Yacoub M, Valeri A, Mangin P, Vallancien G, Cancel-Tassin G, Cussenot O. Differential expression of genes related to androgen and estrogen metabolism in hereditary versus sporadic prostate cancer. Cancer Epidemiol Biomarkers Prev. 2008 Jun;17(6):1505-9. doi: 10.1158/1055-9965.EPI-07-2778. PMID 18559568
- [Background] Thomas G, Jacobs KB, Yeager M, Kraft P, Wacholder S, Orr N, Yu K, Chatterjee N, Welch R, Hutchinson A, Crenshaw A, Cancel-Tassin G, Staats BJ, Wang Z, Gonzalez-Bosquet J, Fang J, Deng X, Berndt SI, Calle EE, Feigelson HS, Thun MJ, Rodriguez C, Albanes D, Virtamo J, Weinstein S, Schumacher FR, Giovannucci E, Willett WC, Cussenot O, Valeri A, Andriole GL, Crawford ED, Tucker M, Gerhard DS, Fraumeni JF Jr, Hoover R, Hayes RB, Hunter DJ, Chanock SJ. Multiple loci identified in a genome-wide association study of prostate cancer. Nat Genet. 2008 Mar;40(3):310-5. doi: 10.1038/ng.91. Epub 2008 Feb 10. PMID 18264096
- [Background] Lou H, Yeager M, Li H, Bosquet JG, Hayes RB, Orr N, Yu K, Hutchinson A, Jacobs KB, Kraft P, Wacholder S, Chatterjee N, Feigelson HS, Thun MJ, Diver WR, Albanes D, Virtamo J, Weinstein S, Ma J, Gaziano JM, Stampfer M, Schumacher FR, Giovannucci E, Cancel-Tassin G, Cussenot O, Valeri A, Andriole GL, Crawford ED, Anderson SK, Tucker M, Hoover RN, Fraumeni JF Jr, Thomas G, Hunter DJ, Dean M, Chanock SJ. Fine mapping and functional analysis of a common variant in MSMB on chromosome 10q11.2 associated with prostate cancer susceptibility. Proc Natl Acad Sci U S A. 2009 May 12;106(19):7933-8. doi: 10.1073/pnas.0902104106. Epub 2009 Apr 21. PMID 19383797
- [Background] Nicolaiew N, Cancel-Tassin G, Azzouzi AR, Grand BL, Mangin P, Cormier L, Fournier G, Giordanella JP, Pouchard M, Escary JL, Valeri A, Cussenot O. Association between estrogen and androgen receptor genes and prostate cancer risk. Eur J Endocrinol. 2009 Jan;160(1):101-6. doi: 10.1530/EJE-08-0321. Epub 2008 Oct 24. PMID 18952763
- [Background] Yeager M, Chatterjee N, Ciampa J, Jacobs KB, Gonzalez-Bosquet J, Hayes RB, Kraft P, Wacholder S, Orr N, Berndt S, Yu K, Hutchinson A, Wang Z, Amundadottir L, Feigelson HS, Thun MJ, Diver WR, Albanes D, Virtamo J, Weinstein S, Schumacher FR, Cancel-Tassin G, Cussenot O, Valeri A, Andriole GL, Crawford ED, Haiman CA, Henderson B, Kolonel L, Le Marchand L, Siddiq A, Riboli E, Key TJ, Kaaks R, Isaacs W, Isaacs S, Wiley KE, Gronberg H, Wiklund F, Stattin P, Xu J, Zheng SL, Sun J, Vatten LJ, Hveem K, Kumle M, Tucker M, Gerhard DS, Hoover RN, Fraumeni JF Jr, Hunter DJ, Thomas G, Chanock SJ. Identification of a new prostate cancer susceptibility locus on chromosome 8q24. Nat Genet. 2009 Oct;41(10):1055-7. doi: 10.1038/ng.444. Epub 2009 Sep 20. PMID 19767755
- [Background] Prokunina-Olsson L, Fu YP, Tang W, Jacobs KB, Hayes RB, Kraft P, Berndt SI, Wacholder S, Yu K, Hutchinson A, Spencer Feigelson H, Thun MJ, Diver WR, Albanes D, Virtamo J, Weinstein S, Schumacher FR, Cancel-Tassin G, Cussenot O, Valeri A, Andriole GL, Crawford ED, Haiman CA, Henderson BE, Kolonel L, Le Marchand L, Siddiq A, Riboli E, Travis R, Kaaks R, Isaacs WB, Isaacs SD, Gronberg H, Wiklund F, Xu J, Vatten LJ, Hveem K, Kumle M, Tucker M, Hoover RN, Fraumeni JF Jr, Hunter DJ, Thomas G, Chatterjee N, Chanock SJ, Yeager M. Refining the prostate cancer genetic association within the JAZF1 gene on chromosome 7p15.2. Cancer Epidemiol Biomarkers Prev. 2010 May;19(5):1349-55. doi: 10.1158/1055-9965.EPI-09-1181. Epub 2010 Apr 20. PMID 20406958
- [Background] Cussenot O, Azzouzi AR, Nicolaiew N, Fromont G, Mangin P, Cormier L, Fournier G, Valeri A, Larre S, Thibault F, Giordanella JP, Pouchard M, Zheng Y, Hamdy FC, Cox A, Cancel-Tassin G. Combination of polymorphisms from genes related to estrogen metabolism and risk of prostate cancers: the hidden face of estrogens. J Clin Oncol. 2007 Aug 20;25(24):3596-602. doi: 10.1200/JCO.2007.11.0908. PMID 17704407
- See also: website from the sponsor which contains a description of the ProGene study and the associated publications — https://cerepp.org/